CLINICAL TRIAL: NCT07013201
Title: A Proof-of-concept Phase 2a, Double-blind, 2-arm Trial to Investigate the Efficacy and Safety of Twice Daily Delgocitinib Cream 20 mg/g Compared With Cream Vehicle During a 16-week Treatment Period in Adult Subjects With Mild to Severe Palmoplantar Pustulosis
Brief Title: A 16-week Trial to Investigate the Efficacy and Safety of Delgocitinib Cream 20 mg/g in Adult Participants With Mild to Severe Palmoplantar Pustulosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0133-2393; 2024-518856-21-00 (EU CTIS Number); U1111-1319-5081 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Palmoplantar Pustulosis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delgocitinib 20 mg/g (Experimental): Participants with mild to severe PPP will receive 20 mg/g of delgocitinib cream twice a day for 16 weeks.
  Interventions: Drug: Delgocitinib cream
- Cream Vehicle (Placebo Comparator): Participants with mild to severe PPP will receive matching vehicle cream twice a day for 16 weeks.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Delgocitinib cream — Topical application
  Arms: Delgocitinib 20 mg/g
Drug: Vehicle cream — Topical application
  Arms: Cream Vehicle

SUMMARY:
The main objective of the study is to evaluate the efficacy of twice daily applications of delgocitinib cream 20 mg/g compared with cream vehicle in the treatment of adult participants with mild to severe palmoplantar pustulosis (PPP). Total study duration for each participants will be approximately 18 weeks, for an approximate total of 9 visits.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent has been obtained prior to any protocol-related procedures.
* Age 18 years or above at the time of informed consent signing.
* Participant is able to comply with clinic visits and trial requirements and procedures, as assessed by the investigator.
* Diagnosis of PPP in accordance with the consensus diagnostic criteria established by European Rare and Severe Psoriasis Expert Network: primary, persistent (>3 months duration), sterile, macroscopically visible pustules on the palms and/or soles, with or without plaque psoriasis elsewhere on the body.
* Confirmed PPP by central evaluation of photographs taken at screening.
* Mild to severe PPP current condition defined by:

  * Disease duration of PPP of >6 months before randomisation.
  * PPP-PGA of at least mild severity (PPP-PGA ≥2) at screening and baseline.
  * PPPASI ≥8 at screening and baseline.
* Presence of ≥5 well-demarcated fresh pustules (white or yellow pustules) in total across all affected areas at screening and baseline.
* Participants with prior experiences of inadequate response with topical corticosteroid(s) (TCS) or for whom TCS are inadvisable, as judged by the investigators.
* A woman of childbearing potential must use an acceptable form of birth control throughout the trial up until the last administration of investigational medicinal product (IMP).

Exclusion Criteria:

* Presence or known history of drug-induced PPP (e.g., a new onset of PPP or an exacerbation of PPP from beta blockers, calcium channel blockers, lithium, or biologic therapy including infliximab, adalimumab, or etanercept).
* Presence of acrodermatitis continua of Hallopeau.
* Active dermatologic condition that could confound the diagnosis of PPP or interfere with assessment of the IMP, as assessed by the investigator.
* Clinically significant infection on the palms or soles.
* Concurrent plaque psoriasis covering >5% of body surface area.
* Clinically significant infection within 4 weeks prior to baseline, which, in the opinion of the investigator, may compromise the safety of the participant in the trial, interfere with evaluation of the IMP, or reduce the participant's ability to participate in the trial. Clinically significant infections are defined as:

  * A systemic infection.
  * A serious skin infection requiring parenteral (intravenous or intramuscular) antibiotics, antiviral, or antifungal medication.
* History of any known primary immunodeficiency disorder, including a positive human immunodeficiency virus test at screening, or the participant taking antiretroviral medications as determined by medical history and/or the participant's verbal report.
* Major surgery within 8 weeks prior to screening or planned in-patient surgery or hospitalisation during the trial period.
* Any documented active or suspected malignancy, or history of malignancy within 5 years prior to screening, except basal cell carcinoma of the skin, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix appropriately treated before the baseline visit.
* Any disorder that is not stable and could:

  * Affect the safety of the participant throughout the trial.
  * Impede the participant's ability to complete the trial. Examples include, but are not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, immunological, and psychiatric disorders, as well as major physical impairment.
* Any clinically significant abnormal finding occurring during the screening period and/or observed at the baseline visit that may put the participant at risk due to their participation in the trial or could influence the participant's ability to complete the trial.
* Positive hepatitis B surface antigen and/or hepatitis B core antibody and positive hepatitis B virus DNA (participants who have tested positive for hepatitis B core antibody are eligible if tests for hepatitis B surface antigen and hepatitis B virus DNA are negative) or positive hepatitis C virus antibody serology confirmed by hepatitis C virus RNA at screening.
* Known or suspected hypersensitivity to any component(s) of the IMP.
* Current or recent chronic alcohol or drug abuse, or any other condition associated with poor compliance as judged by the investigator.
* Women who are pregnant or lactating.
* Systemic treatment within 4 weeks prior to baseline with immunosuppressive drugs (e.g., methotrexate, cyclosporine, azathioprine), immunomodulating drugs, retinoids (e.g., acitretin), tyrosine kinase inhibitors, phosphodiesterase-4 inhibitors, or corticosteroids (steroid eye drops and inhaled or intranasal steroids in the doses recommended in the product prescribing information for the treatment of allergic conjunctivitis, asthma, or rhinitis are allowed).
* Use of tanning beds or phototherapy (e.g., ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen ultraviolet A [PUVA]) on the palms or soles within 4 weeks prior to baseline.
* Use of systemic or topical janus kinase inhibitors (including delgocitinib/LEO 124249) within 4 weeks prior to baseline.
* Cutaneously applied treatment with immunomodulators (e.g., phosphodiesterase-4 [PDE-4] inhibitors, pimecrolimus, tacrolimus, tapinarof, vitamin D3 derivatives) or TCS on the palms or soles within 2 weeks prior to baseline.
* Use of systemic antibiotics or cutaneously applied antibiotics on the palms or soles within 2 weeks prior to baseline.
* Other transdermal or cutaneously applied therapy on the palms or soles (except for the use of the participant's own non-medicated emollients) within 1 week prior to baseline.
* Cutaneously applied treatments in regions other than the palms or soles, which could interfere with clinical trial evaluations or pose a safety concern (excluding treatments for psoriasis patches or other non-exclusionary skin conditions, if needed) within 1 week prior to baseline.
* Treatment with any marketed biological therapy or investigational biologic agents:

  * Any cell-depleting agents, including but not limited to rituximab: within 6 months prior to baseline, or until lymphocyte count returns to normal, whichever is longer.
  * Other biologics, including but not limited to secukinumab, ustekinumab, tildrakizumab, ixekizumab, risankizumab, guselkumab, and tumour necrosis factor (TNF)-alpha inhibitors: within 3 months or 5 half-lives, whichever is longer, prior to baseline.
* Treatment with any non-marketed drug substance (i.e., an agent that has not yet been made available for clinical use following registration) within the last 4 weeks prior to baseline or 5 half-lives, whichever is longer.
* Current participation in any other interventional clinical trial.
* Previously randomised in this clinical trial.
* Previously randomised in a clinical trial with delgocitinib.
* Employees of the trial site, or any other individuals directly involved with the planning or conduct of the trial, or immediate family members of such individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving at Least 75% Improvement in PPP Area and Severity Index (PPPASI) Score from Baseline (PPPASI-75) at Week 16 | Baseline to Week 16

SECONDARY OUTCOMES:
Number of Participants with PPP-Physician Global Assessment (PGA) Score of 0 or 1 with at Least a 2-step Improvement from Baseline at Week 16 | Baseline to Week 16
Change in the Overall Number of Fresh Pustules From Baseline to Week 16 | Baseline to Week 16
Number of Participants with a ≥1-point Reduction in PPP-PGA Score From Baseline to Week 16 | Baseline to Week 16
Number of Participants with a ≥2-point Reduction in PPP-PGA Score From Baseline to Week 16 | Baseline to Week 16
Change in PPPASI Score From Baseline to Week 16 | Baseline to Week 16
Percentage Change in PPPASI Score From Baseline to Week 16 | Baseline to Week 16
Number of Participants Achieving PPPASI-50 at Week 16 | Week 16
Number of Participants Achieving PPPASI-90 at Week 16 | Week 16
Change from Baseline to Week 16 in PPP-symptoms assessment (SA) Score | Baseline to Week 16
Percentage Change in PPP-SA Score from Baseline to Week 16 | Baseline to Week 16
Change from Baseline to Week 16 in PPP-SA Itch Score for the Hands | Baseline to Week 16
Change from Baseline to Week 16 in PPP-SA Itch Score for the Feet | Baseline to Week 16
Change from Baseline to Week 16 in PPP-SA Pain Score for the Hands | Baseline to Week 16
Change from Baseline to Week 16 in PPP-SA Pain Score for the Feet | Baseline to Week 16
Change in Fresh Pustules at Weeks 1, 2, 4, 8, and 12 | Baseline to Week 12
Number of Fresh Pustules Overall at Weeks 1, 2, 4, 8, 12, and 16 | Baseline to Week 16
Number of Participants who Experienced Treatment-emergent Adverse Events (TEAEs) | Baseline to Week 18
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurred after the participant received study treatment. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration were recorded as TEAEs. A serious TEAE is any untoward medical occurrence in a clinical study participant after first dose irrespective of a causal relationship with the study treatment(s) that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
Number of Participants with a ≥4-point Reduction in Dermatology Life Quality Index (DQLI) Score From Baseline to Week 16 | Baseline to Week 16
Change from Baseline to Week 16 in DLQI Score | Baseline to Week 16
Percentage Change from Baseline to Week 16 in DLQI Score | Baseline to Week 16
Change from Baseline to Week 16 in PPP-Impact Assessment (IA) Score | Baseline to Week 16
Percentage Change from Baseline to Week 16 in PPP-IA Score | Baseline to Week 16
Change in Work Productivity and Activity (WPAI) PPP Absenteeism Score from Baseline to Week 16 | Baseline to Week 16
Change in Work WPAI:PPP Presenteeism Score from Baseline to Week 16 | Baseline to Week 16
Change in WPAI:PPP work Productivity Score from Baseline to Week 16 | Baseline to Week 16
Change in WPAI:PPP Activity Impairment Score from Baseline to Week 16 | Baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (30):
- United States (7):
  - LEO Pharma Investigational Site, Fountain Valley, California
  - LEO Pharma Investigational Site, Douglasville, Georgia
  - LEO Pharma Investigational Site, West Bloomfield, Michigan
  - LEO Pharma Investigational Site, Elmhurst, New York
  - LEO Pharma Investigation Site, Mayfield Heights, Ohio
  - LEO Pharma Investigational Site, Portland, Oregon
  - LEO Pharma Investigational Site, Philadelphia, Pennsylvania
- Canada (7):
  - LEO Pharma Investigational Site, Surrey, British Columbia
  - LEO Pharma Investigational Site, Winnipeg, Manitoba
  - LEO Pharma Investigational Site, Fredericton, New Brunswick
  - LEO Pharma Investigational Site, Hamilton, Ontario
  - LEO Pharma Investigational Site, Markham, Ontario
  - LEO Pharma Investigational Site, Waterloo, Ontario
  - LEO Pharma Investigational Site, Montreal, Quebec
- Germany (8):
  - LEO Pharma Investigational Site, Bad Bentheim
  - LEO Pharma Investigational Site, Dresden
  - LEO Pharma Investigational Site, Kiel
  - LEO Pharma Investigational Site, Lübeck
  - LEO Pharma Investigational Site, Manheim
  - LEO Pharma Investigational Site, Münster
  - LEO Pharma Investigational Site, Osnabrück
  - LEO Pharma Investigational Site, Witten
- Poland (7):
  - LEO Pharma Investigational Site, Bialystok
  - LEO Pharma Investigational Site, Iwonicz-Zdrój
  - LEO Pharma Investigational Site, Lodz
  - LEO Pharma Investigational Site, Lublin
  - LEO Pharma Investigational Site, Rzeszów
  - LEO Pharma Investigational Site, Warsaw
  - LEO Pharma Investigational Site, Wroclaw
- LEO Pharma Investigational Site, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No